CLINICAL TRIAL: NCT02944149
Title: Safety of Minilaparotomy Provided by Trained Clinical Officers and Assistant Medical Officers: a Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EngenderHealth (Other)
Collaborators: Tanzania Ministry of Health, Community Development, Gender, Elders, and Children (Unknown); Association of Gynaecologists and Obstetricians of Tanzania (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TAN-42
Record Dates: First submitted 2016-10-14; First posted 2016-10-25 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Sterilization, Tubal
MeSH Terms: interventions — Sterilization, Reproductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- assistant medical officer (AMO) (Active Comparator): Assistant medical officers (AMO) are currently allowed to provide tubal ligation by minilaparotomy, however government regulations do not allow clinical officers (COs) to provide this service.
  Interventions: Procedure: tubal ligation by minilaparotomy
- clinical officer (CO) (Experimental): Experimental: clinical officer (CO) In Tanzania, COs are mid-level providers who offer diagnosis, treatment, and minor surgeries. They are more common in rural areas than medical officers (MOs) and assistant medical officers (AMOs) and are generally considered capable of performing minor surgery. Almost all facilities in Tanzania are understaffed, but COs vastly outnumber MOs and AMOs. COs are more prevalent in poorer and/or rural areas than other higher level cadres; thus, task-shifting to COs would increase access to tubal ligation by minilaparotomy for many women who are most in need.
  Interventions: Procedure: tubal ligation by minilaparotomy

INTERVENTIONS:
Procedure: tubal ligation by minilaparotomy — Tubal ligation will be performed by minilaparotomy as per the Tanzanian government standards, with the standard family planning counseling and minilaparotomy surgical protocols used by the government being followed during the study.
  Other Names: female sterilization

SUMMARY:
The study is a non-inferiority randomized controlled trial (RCT) that aims to demonstrate that tubal ligations by minilaparotomy (ML) conducted by trained clinical officers (COs) are no less safe as compared to those conducted by assistant medical officers (AMOs) in Tanzania. Participants will be randomized in a one to one ratio to ML by a CO and ML by an AMO. In addition to the screening and enrollment/ML visit, there will be three scheduled follow-up visits at 3, 7 and 42 days post-surgery.

DETAILED DESCRIPTION:
The primary objective is to establish whether the safety of ML provided by trained COs is not inferior to the safety of ML provided by trained AMOs, as measured by rates of major adverse events (AEs) among women undergoing ML. The primary outcome is safety, defined by the overall rate of major AEs following ML. The investigators will address the primary objective by comparing the rate of major AEs observed following MLs conducted by COs vs. AMOs during the ML procedure and through 42 days follow-up. This study will be conducted among 1,970 women 18 years of age and older presenting at study sites for ML surgery. The duration of a woman's participation in the study is expected to be 6 weeks, unless additional follow-up beyond 42 days is clinically indicated due to complications or for other reasons. The study will be conducted in Arusha Region in northern Tanzania. The following health facilities will serve as study sites: Daraja Health Centre, Karatu Hospital, Kaloleni Health Centre, Levolosi Urban Health Centre, Longido Health Centre, Monduli Hospital, and Mto wa Mbu Health Centre.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older;
* Requested and consented to female sterilization AND additionally freely consents to participate in the study and signs a study informed consent form;
* Is sound of mind, in good general health and deemed suitable to undergo female sterilization by ML in accordance with the Tanzania government guidelines;
* Able to understand study procedures and requirements of study participation;
* Agrees to return to the study site for the full schedule of follow-up visits after her ML procedure;
* Agrees to provide the study staff with an address, phone number, close relative, and/or other locator information while participating in the research study.

Exclusion Criteria:

* Pregnancy
* Between 8 and 42 days postpartum or postabortion
* Known allergy or sensitivity to lidocaine or other local anesthesia
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid
* Previous abdominal or pelvic surgery
* Local skin infection near area where incision will be made
* Coagulation disorder
* Hypertension (properly taken measurements; systolic ≥ 160 or diastolic ≥ 100 mm Hg)
* Acute deep venous thrombosis/pulmonary embolism
* Current ischemic heart disease
* Unexplained vaginal bleeding
* Malignant gestational trophoblastic disease
* Cervical, endometrial and/or ovarian cancer
* Pelvic inflammatory disease (current or within the last three months)
* Current purulent cervicitis, chlamydial infection and/or gonorrhea
* Current symptomatic gall bladder disease
* Active viral hepatitis
* Severe anemia (irrespective of type or etiology)
* Tuberculosis of pelvic organs
* Acute bronchitis or pneumonia
* Systematic infection or gastroenteritis
* Currently participating in another biomedical research study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1970 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safety: safety is defined by the overall rate of major adverse events (AEs) during and after the procedure. Rates of major AEs observed during and after procedures conducted by COs vs. AMOs will be compared. | During the minilaparotomy procedure and through 42 days follow-up

SECONDARY OUTCOMES:
Performance | During the minilaparotomy procedure
  Performance assessed by (e.g., procedure times, difficulties performing the procedure, inability to complete the procedure, need for assistance to complete the procedure, maximum reported pain experienced by the participant during the procedure) between procedures performed by COs and AMOs will be compared
Participant satisfaction | During the minilaparotomy procedure and through 42 days follow-up
  Participant satisfaction with the minilaparotomy experience conducted by COs and AMOs will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Barone, DVM, MS, Principal Investigator — EngenderHealth
Locations (7):
- Tanzania (7):
  - Daraja Health Centre, Arusha, Arusha
  - Kaloleni Health Centre, Arusha, Arusha
  - Levolosi Health Centre, Arusha, Arusha
  - Karatu Lutheran Hospital, Kiratu, Arusha
  - Longido Health Centre, Longido, Arusha
  - Monduli District Hospital, Monduli, Arusha
  - Mto Wa Mbu Health Center, Monduli, Arusha

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barone MA, Mbuguni Z, Achola JO, Almeida A, Cordero C, Kanama J, Marquina A, Muganyizi P, Mwanga J, Ouma D, Shannon C, Tibyehabwa L. Safety of Tubal Occlusion by Minilaparotomy Provided by Trained Clinical Officers Versus Assistant Medical Officers in Tanzania: A Randomized, Controlled, Noninferiority Trial. Glob Health Sci Pract. 2018 Oct 4;6(3):484-499. doi: 10.9745/GHSP-D-18-00108. Print 2018 Oct 3. PMID 30120168
- [Derived] Barone MA, Mbuguni Z, Achola JO, Cordero C, Kanama J, Muganyizi PS, Mwanga J, Shannon C, Tibyehabwa L. Safety of tubal ligation by minilaparotomy provided by clinical officers versus assistant medical officers: study protocol for a noninferiority randomized controlled trial in Tanzanian women. Trials. 2017 Oct 26;18(1):499. doi: 10.1186/s13063-017-2235-6. PMID 29073928